CLINICAL TRIAL: NCT06981546
Title: Modeling Clinical Outcomes in Gambling Addiction
Acronym: MOGADOR
Status: Not yet recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0270; 2024-A01805-42 (Other: ID-RCB)
Record Dates: First submitted 2025-05-05; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Gambling Disorder
Keywords: Gambling disorders; Modeling outcomes; Socio-demographic Characteristics; Clinical psychiatric profiles
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with gambling disorder: OGADOR will focus exclusively on patients with DSM-5 criteria for gambling disorder and on demand for medical care. In this study psychiatric and addictological comorbidities, frequent in such a cohort, will constitute a specific inclusion factor, key characteristic leading an analysis of the impact on the patient prognosis.

SUMMARY:
Gambling disorder (GD) is recognized as an addictive disorder. Financial consequences of GD are often dramatic, inducing professional, familial, legal and medical repercussions and particularly mental health consequences.

MOGADOR is a longitudinal, multicentric, prospective, prognostic study, which aims to identify factors predicting the evolution of french patients with GD in care centers particularly involved in the management of GD. The main goal will focus on evolution of DSM-5 (Diagnostic and Statistical Manual of Mental Disorder 5th edition) GD criteria during the first year of follow-up. The prognostic factors will be collected at base-line and they will be considered to influence the long-term prognosis of patients.

For patients suffering of GD, our main hypothesis is that initial factors like individual socio-demographic characteristics, clinical psychiatric profiles, addiction comorbidities, and behaviour are associated with the clinical prognosis (total remission of DSM-5 criteria of GD at 12 months).

MOGADOR will be the first study, aiming to model prognostic aspects of GB in populations specially monitored for this disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, over 18 years old, consulting in one of the participating centers.
* DSM-5 criteria for gambling disorder at inclusion: at least 4 criteria present in the 12 months preceding the study.
* First treatment for gambling disorder or no treatment in the last 6 months (initiation or re-initiation of care).

Exclusion Criteria:

* Unable to be reached by phone.
* Unable to use the internet.
* Patient under antiparkinsonian treatment of the dopaminergic family.
* Being treated with a drug that may trigger/increase symptoms of gambling disorder (e.g. dopamine agonist).
* Subject under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 268 patients with gambling disorder according to DSM-5 criteria newly managed in one of the participating centers or who had an interruption in management of more than 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 268 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Partial remission of gambling disorder at 12 months (strictly less than 4 DSM-5 criteria) | DSM-5 criteria assessment will be conducted at 9 and 12 months after inclusion.
  Assessment of DSM-5 criteria will be performed by the clinician, and by a previously trained CRA if clinical follow-up is discontinued.
modeling prognostic factors | at inclusion visit.
  The prognostic factors, studied will be: number of initial DSM-5 criteria, gender, age, marital status, housing, employment status, socioeconomic level, time spent gambling, impulsivity, type of gambling, location of gambling, and also the factor with the strongest association in univariate analysis among the following factors:
  * Depression (PHQ scale),
  * Anxiety (GAD scale),
  * Quality of life (SF-36 scale).

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - Hôpital Jen Minjoz, CHU de Besançon, Besançon
  - Service Universitaire d'Addictologie de Lyon (SUAL), CH Le Vinatier, Bron
  - Service Universitaire d'Addictologie de Lyon (SUAL), Groupement Hospitalier Est, Bron
  - Service Universitaire d'Addictologie, CHU de Clermont-Ferrand, Clermont-Ferrand
  - Name of location * Service d'Addictologie, Groupe Hospitalier Seclin Carvin, Lille
  - Centre Expert Régional du Jeu Pathologique (CERJeP Limousin), Limoges
  - Service Universitaire d'Addictologie, CHU de Nîmes, Nîmes
  - Assistance Publique des Hôpitaux de Paris, Hôpital Marmottan, Paris
  - Hôpital de Bellevue, CHU de St-Etienne, Saint-Etienne